CLINICAL TRIAL: NCT05292131
Title: An Open-Label, Randomized, Parallel-Group, Single-Dose Bioequivalence Study of Bimekizumab Given as 1x2mL or 2x1mL Subcutaneous Injection Using an Autoinjector in Healthy Study Participants
Brief Title: A Bioequivalence Study of Bimekizumab Given as 1x2mL or 2x1mL Subcutaneous Injection Using an Autoinjector in Healthy Study Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: UCB Biopharma SRL (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: UP0119
Record Dates: First submitted 2022-03-14; First posted 2022-03-23 (Actual); Results first posted 2025-04-10 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-03

CONDITIONS: Healthy Study Participants
Keywords: UCB4940; BKZ; bimekizumab; Bioequivalence; Auto-injector; Healthy study participants
MeSH Terms: interventions — bimekizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Test (Experimental): Study participants randomized to this arm will receive bimekizumab (BKZ) administered subcutaneously with bimekizumab-AI-2mL presentation (test).
  Interventions: Drug: bimekizumab
- Reference (Other): Study participants randomized to this arm will receive bimekizumab (BKZ) administered subcutaneously with bimekizumab-AI-1x2mL presentation (reference).
  Interventions: Drug: bimekizumab

INTERVENTIONS:
Drug: bimekizumab — Study participants will receive a single dose of bimekizumab (BKZ) administered subcutaneously in the Treatment Period.
  Other Names: BKZ; UCB4940

SUMMARY:
The purpose of the study is to compare the pharmacokinetics (PK), safety and tolerability of a single subcutaneous (sc) dose of bimekizumab (BKZ) when administered using bimekizumab-autoinjector (AI)-2mL presentation versus bimekizumab-AI-2x1mL presentation in healthy study participants.

ELIGIBILITY:
Inclusion Criteria:

* Study participant must be ≥18 years and ≤65 years of age inclusive, at the time of signing the informed consent
* Study participants who are overtly healthy as determined by medical evaluation including medical history, physical examination, vital signs, 12-lead electrocardiogram (ECG), and laboratory tests, during the Screening Period and on admission
* Study participant has a body temperature between 35.0°C and 37.5°C, inclusive, at Screening and on admission
* Body weight minimum of 50 kg for male and 45 kg for female study participants and a maximum of 100 kg for all study participants, and body mass index (BMI) within the range 18 to 32 kg/m^2 (inclusive) at the Screening Visit
* Male or female. Contraception guidelines (as per the standard UCB contraceptive guideline) will be applicable.

Exclusion Criteria:

* Study participant has a known hypersensitivity to any components of the bimekizumab (and/or an investigational device) as stated in this protocol
* Study participant has an active infection or history of infections as follows:
* Any active infection (except common cold) within 14 days prior to Screening Visit
* A serious infection, defined as requiring hospitalization or iv anti-infectives within 2 months prior to the Screening Visit
* A history of opportunistic, recurrent, or chronic infections that, in the opinion of the Investigator, might cause this study to be detrimental to the study participant. Opportunistic infections are infections caused by uncommon pathogens (eg, pneumocystis jirovecii, cryptococcosis) or unusually severe infections caused by common pathogens (eg, cytomegalovirus, herpes zoster)
* Study participant has a history of a positive TB test or evidence of possible TB or latent TB infection at Screening Visit. Refer to Tuberculosis Detection Procedure Guideline for details regarding TB infection status, detection procedures, and the related exclusion criteria
* Study participants receiving any live (includes attenuated) vaccination within the 8 weeks prior to the Screening Visit (eg, inactivated influenza and pneumococcal vaccines are allowed, but nasal influenza vaccination is not permitted). Live vaccines are not allowed during the study or for 20 weeks after the last dose of the investigational medicinal product (IMP)
* Study participant has previously participated in this study or a study participant has previously been assigned to bimekuzimab treatment in any other study
* Exposure to 3 or more new chemical entities within 12 months prior to dosing
* Current enrollment or past participation within the last 30 days before signing the informed consent form (ICF) in any other clinical study involving an investigational study intervention or any other type of medical research
* Study participant has concurrent acute or chronic viral hepatitis B or C or human immunodeficiency virus (HIV) infection. Study participants who have evidence of, or tested positive for hepatitis B or hepatitis C are excluded
* Study participant has made a blood donation of a blood loss of more than 400 mL of blood or blood products within 90 days prior to admission (Day -1) or plans to donate blood during the study
* Female study participant who is pregnant, or plans to become pregnant during the study, or lactating, or sexually active with childbearing potential who is not using a medically accepted birth control method
* Study participant has an alcohol consumption of more than 21 units (males) or 14 units (females) of alcohol per week (1 unit of alcohol is equivalent to 12.5 mL ethanol at room temperature)
* Study participant tests positive for alcohol or drugs (urine test) at Screening or Day -1
* Vulnerable study participants (eg, participants kept in detention, protected adults under guardianship or trusteeship, and soldiers or participants committed to an institution by governmental or juridical order), employees of the Sponsor or the contract research organization (CRO) with direct involvement in the proposed study or other studies under the direction of the Investigator or the CRO, as well as family members of the employees or the Investigator
* Study participant has a positive test result for severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) in real-time reverse transcriptase polymerase chain reaction (RT-PCR) on the admission sample
* Study participant has clinical signs and symptoms consistent with COVID-19, eg fever, dry cough, dyspnea, sore throat, fatigue, or confirmed infection by appropriate laboratory test within the previous 14 days prior to Screening or on admission
* Study participant who had severe course of COVID-19 (ie, hospitalization, extracorporal membrane oxygenation, mechanically ventilated)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2022-03-17 (Actual); Primary Completion 2023-01-09 (Actual); Study Completion 2023-01-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — 001 844 599 2273
Locations (2):
- UP0119 2, Glendale, California, United States
- UP0119 1, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No
Data from Phase 1 trials in Healthy Volunteers is outside of UCB's data sharing policy and is unavailable for sharing.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study started to enroll participants in March 2022 and concluded in January 2023.
Pre-assignment Details: The Participant Flow refers to the Safety Set (SS). The SS consisted of all study participants who randomized and received full or partial investigational medicinal product (IMP) according to the treatment the study participants actually received.
Groups:
- Bimekizumab-AI-2mL (Test): Participants received a single dose of bimekizumab 320 mg (1x320 mg) administered as a subcutaneous injection using a 2 mL auto-injector (AI) on Day 1 of the study.
- Bimekizumab-AI-2x1mL (Reference): Participants received a single dose of bimekizumab 320 mg (2x160 mg) administered as a subcutaneous injection using 2x1 mL AI on Day 1 of the study.
Period: Overall Study
Arm/Group | Bimekizumab-AI-2mL (Test) | Bimekizumab-AI-2x1mL (Reference)
Started | 60 | 61
Completed | 59 | 59
Not Completed | 1 | 2
Not completed — Lost to Follow-up | 1 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: Baseline characteristics refer to the SS which consisted of all study participants randomized and received full or partial IMP according to the treatment the participants actually received.
Groups:
- Total: Total of all reporting groups
Arm/Group | Bimekizumab-AI-2mL (Test) | Bimekizumab-AI-2x1mL (Reference) | Total
Number analyzed (Participants) | 60 | 61 | 121
Age, Continuous [Mean (Standard Deviation); unit: Years] | 45.6 (11.7) | 44.8 (11.3) | 45.2 (11.5)
Age, Customized [Count of Participants; unit: Participants]
  18 - <65 yrs | 60 | 59 | 119
  65 - <85 yrs | 0 | 2 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 24 | 48
  Male | 36 | 37 | 73
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 4 | 3 | 7
  Black or African American | 4 | 6 | 10
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  White | 50 | 50 | 100
  Other or Mixed | 1 | 2 | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 12 | 24
  Not Hispanic or Latino | 48 | 49 | 97

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to Infinity (AUC) for a Single Dose Bimekizumab (BKZ)
Description: AUC is the area under the plasma concentration-time curve from time 0 (Day 1 predose) to infinity.
Time Frame: Baseline (Day 1 predose) at predefined time points (up to Day 140)
Population: The Pharmacokinetic Set (PKS) was a subset of the SS, consisted of those study participants that received at least 1 total dose of IMP and had at least 1 observable pharmacokinetic measurement and who had no important protocol deviations affecting pharmacokinetics (PK) during the whole study phase. Number of participants analyzed included those participants who were evaluable for the assessment.
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: days*micrograms/milliliter (days*ug/mL)
Arm/Group | Bimekizumab-AI-2mL (Test) | Bimekizumab-AI-2x1mL (Reference)
Number analyzed (Participants) | 60 | 59
days*micrograms/milliliter (days*ug/mL) | 1223 [1146.1 to 1306.1] | 1255 [1174.2 to 1341.1]
Statistical Analysis 1: Comparison: Bimekizumab-AI-2mL (Test) vs Bimekizumab-AI-2x1mL (Reference); Test type: Equivalence — Bioequivalence (BE) was concluded if the 90% CIs for the ratio of the respective comparison are fully included in the acceptance range from 0.8 to 1.25 for AUC; Geometric Mean Ratio (percentage [%]) = 97.50, 90% CI 2-sided [90.20 to 105.40]

2. Primary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to Last Quantifiable Concentration (AUC0-t) for a Single Dose Bimekizumab (BKZ)
Description: AUC0-t is the area under the plasma concentration-time curve from time zero (Day 1 predose) to the last quantifiable concentration.
Time Frame: From Baseline (Day 1 predose) at predefined time points to the last quantifiable concentration (Day 140)
Population: The PKS was a subset of the SS, consisted of those study participants that received at least 1 total dose of IMP and had at least 1 observable pharmacokinetic measurement and who had no important protocol deviations affecting PK during the whole study phase. Number of participants analyzed included those participants who were evaluable for the assessment.
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: day*ug/mL
Arm/Group | Bimekizumab-AI-2mL (Test) | Bimekizumab-AI-2x1mL (Reference)
Number analyzed (Participants) | 60 | 59
day*ug/mL | 1186 [1114.7 to 1262.9] | 1223 [1147.3 to 1302.6]
Statistical Analysis 1: Comparison: Bimekizumab-AI-2mL (Test) vs Bimekizumab-AI-2x1mL (Reference); Test type: Equivalence — BE was concluded if the 90% CIs for the ratio of the respective comparison are fully included in the acceptance range from 0.8 to 1.25 for AUC0-t; Geometric Mean Ratio (%) = 97.05, 90% CI 2-sided [90.10 to 104.55]

3. Primary Outcome: Maximum Plasma Concentration (Cmax) for a Single Dose Bimekizumab (BKZ)
Description: Cmax is a maximum observed plasma concentration.
Time Frame: From Baseline (Day 1 predose) at predefined time points (up to Day 140)
Population: as for outcome 2
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: micrograms/milliliter (ug/mL)
Arm/Group | Bimekizumab-AI-2mL (Test) | Bimekizumab-AI-2x1mL (Reference)
Number analyzed (Participants) | 60 | 60
micrograms/milliliter (ug/mL) | 35.17 [32.8 to 37.7] | 36.55 [34.1 to 39.2]
Statistical Analysis 1: Comparison: Bimekizumab-AI-2mL (Test) vs Bimekizumab-AI-2x1mL (Reference); Test type: Equivalence — BE was concluded if the 90% CIs for the ratio of the respective comparison are fully included in the acceptance range from 0.8 to 1.25 for Cmax; Geometric Mean Ratio (%) = 96.21, 90% CI 2-sided [88.60 to 104.47]

4. Secondary Outcome: Percentage of Participants With at Least One Treatment-emergent Adverse Event (TEAE) From Baseline to End of Safety Follow-Up
Description: An AE is any untoward medical occurrence in a patient or clinical study participant administered a pharmaceutical product, which does not necessarily have a causal relationship with this treatment. An AE could therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product. TEAEs are defined as AEs not present prior to the administration of IMP or any unresolved event already present before administration of IMP that worsens in intensity following exposure to study treatment.
Time Frame: From Baseline (Day 1) to end of Safety Follow-Up (up to Day 140)
Population: The SS consisted of all study participants who randomized and received full or partial IMP according to the treatment the study participants actually received.
Measure: Number; unit: percentage of participants
Arm/Group | Bimekizumab-AI-2mL (Test) | Bimekizumab-AI-2x1mL (Reference)
Number analyzed (Participants) | 60 | 61
percentage of participants | 43.3 | 49.2

5. Secondary Outcome: Percentage of Participants With at Least One Treatment-emergent Serious Adverse Event (SAE) From Baseline to End of Safety Follow-Up
Description: A SAE is defined as any untoward medical occurrence that at any dose: a. Results in death, b. Is life-threatening, c. Requires inpatient hospitalization or prolongation of existing hospitalization, d. Results in persistent disability/incapacity, e. Is a congenital anomaly/ birth defect, f. Is an important medical event which based on appropriate medical judgment, jeopardized the study participant and required medical or surgical intervention to prevent any of the above.
Time Frame: From Baseline (Day 1) to end of Safety Follow-Up (up to Day 140)
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Bimekizumab-AI-2mL (Test) | Bimekizumab-AI-2x1mL (Reference)
Number analyzed (Participants) | 60 | 61
percentage of participants | 0 | 0

6. Secondary Outcome: Apparent Terminal Half-life (t1/2)
Description: Apparent terminal half-life as determined via linear regression (slope=-lamdbaz) of the natural log (ln) concentration versus time, for data points in the terminal phase of the concentration time curve (ln2/lambdaz).
Time Frame: From Baseline (Day 1 predose) at predefined time points (up to Day 140)
Population: as for outcome 2
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: days
Arm/Group | Bimekizumab-AI-2mL (Test) | Bimekizumab-AI-2x1mL (Reference)
Number analyzed (Participants) | 60 | 59
days | 24.65 [23.2 to 26.2] | 24.38 [22.9 to 25.9]
Statistical Analysis 1: Comparison: Bimekizumab-AI-2mL (Test) vs Bimekizumab-AI-2x1mL (Reference); Test type: Equivalence — BE was concluded if the 90% CIs for the ratio of the respective comparison are fully included in the acceptance range from 0.8 to 1.25 for t½; Geometric Mean Ratio (%) = 101.13, 90% CI 2-sided [94.18 to 108.59]

7. Secondary Outcome: Time of Occurrence of the Maximum Observed Concentration (Tmax) of a Single Dose Bimekizumab (BKZ)
Description: tmax is the time to reach maximum plasma concentration.
Time Frame: From Baseline (Day 1 predose) at predefined time points (up to Day 140)
Population: as for outcome 2
Measure: Median (Full Range); unit: day
Arm/Group | Bimekizumab-AI-2mL (Test) | Bimekizumab-AI-2x1mL (Reference)
Number analyzed (Participants) | 60 | 60
day | 6.962 [2.96 to 12.0] | 5.979 [2.00 to 21.0]
Statistical Analysis 1: Comparison: Bimekizumab-AI-2mL (Test) vs Bimekizumab-AI-2x1mL (Reference); Test type: Equivalence — The point estimate and the 90% CI for the median treatment differences for tmax was computed according to the Hodges-Lehmann's method; Hodges-Lehman Estimate = 0.4897, 90% CI 2-sided [-0.0073 to 0.9567]

ADVERSE EVENTS:
Time Frame: From Baseline (Day 1) to end of Safety Follow-Up (up to Day 140)
Description: TEAEs are defined as AEs not present prior to the administration of IMP or any unresolved event already present before administration of IMP that worsens in intensity following exposure to study treatment. The SS consisted of all study participants who randomized and received full or partial IMP according to the treatment the study participants actually received.
Arm/Group | Bimekizumab-AI-2mL (Test) | Bimekizumab-AI-2x1mL (Reference)
All-Cause Mortality (participants affected / at risk) | 0/60 | 0/61
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/61
Other Adverse Events (participants affected / at risk) | 11/60 | 16/61
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bimekizumab-AI-2mL (Test) (N=60) | Bimekizumab-AI-2x1mL (Reference) (N=61)
Fatigue (General disorders) | 1 (2) | 4 (4)
Nasopharyngitis (Infections and infestations) | 4 (4) | 7 (8)
Headache (Nervous system disorders) | 8 (14) | 8 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2022-03-21): https://cdn.clinicaltrials.gov/large-docs/31/NCT05292131/Prot_000.pdf
  • Statistical Analysis Plan (2023-02-02): https://cdn.clinicaltrials.gov/large-docs/31/NCT05292131/SAP_001.pdf